CLINICAL TRIAL: NCT03131830
Title: Individual Choice of Delivery Mode - A Prospective Study Using Online Surveys
Brief Title: Individual Choice of Delivery Mode
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: DECISION
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2017-04

CONDITIONS: Delivery Mode

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Staff of the University Clinic of Tuebingen: Online-based questionnaire
  Interventions: Other: Online-based questionnaire
- Participants of the 9th German Urogynecological Congress: Online-based questionnaire
  Interventions: Other: Online-based questionnaire
- All members of the German Society of Obsetrics and Gynecology: Online-based questionnaire
  Interventions: Other: Online-based questionnaire
- Pregnant women from Tübingen and Heidelberg: Online-based questionnaire
  Interventions: Other: Online-based questionnaire

INTERVENTIONS:
Other: Online-based questionnaire — Participants receive a web-link to a questionnaire, which is active for 3 months

SUMMARY:
The primary aim of the study is to investigate personal attitudes regarding mode of delivery among both medical health care professionals and non-professionals. The investigators are also investigating whether providing detailed information that might influence one's decision regarding mode of delivery (such as education on pelvic floor disorders or advantages or disadvantages of epidural anaesthesia) will change participants´ opinion how to determine their preferred mode of delivery.

DETAILED DESCRIPTION:
The choice of delivery mode is an individual decision that is affected by personal opinions and feelings about what might be best for one's own body and child. Increasing awareness about the risks of vaginal delivery has led to an increasing rate of cesearean delivery on maternal request.

The primary aim of the study is to investigate personal attitudes regarding mode of delivery among both medical health care professionals and non-professionals. The investigators are also investigating whether providing detailed information that might influence one's decision regarding mode of delivery (such as education on pelvic floor disorders or advantages or disadvantages of epidural anaesthesia) will change participants´ opinion how to determine their preferred mode of delivery.

A secondary aim of the survey is to gather information about personal attitudes regarding:

* epidural anaesthesia for pain relief during delivery
* systems of risk stratification
* postnatal recovery exercises The data will be acquired with an online questionnaire designed for this study. There will be two groups in this study. The first group ("medical professionals") consists of gynecologists with either subspecialization (urogynecology , fetal and maternal medicine, obstetrics, other) and other non-OB/GYN health care providers and medical staff, regardless whether they are nurses, medical assistants, physicians, physiotherapists, midwifes, administration staff. The group of "non-professionals" consists of women who are currently pregnant, and are not healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* able to fill out a questionnaire

Exclusion Criteria:

* minor people

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There will be two groups in this study. The first group ("medical professionals") consists of gynecologists with either subspecialization (urogynecology , fetal and maternal medicine, obstetrics, other) and other non-OB/GYN health care providers and medical staff, regardless whether they are nurses, medical assistants, physicians, physiotherapists, midwifes, administration staff. The group of "non-professionals" consists of women who are currently pregnant, and are not healthcare professionals.
  Inclusion Criteria:
  Participants in the "medical professionals" group can be from either gender, over age 18, currently working in the medical profession and have sufficient understanding of the German language in order to be able to fill out the questionnaire.
  The "non-professionals" are pregnant females over age 18 with sufficient understanding of the German language in order to be able to fill out the questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 2605 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Delivery mode | 3 months
  Choice of delivery mode

CONTACTS AND LOCATIONS:
Locations (1):
- University Women's Hospital, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No